CLINICAL TRIAL: NCT06284226
Title: An Exploratory Clinical Study to Evaluate the Safety and Efficacy of NK Cells (Combined With Standard Therapy) in the Treatment of Solid Tumor Patients
Acronym: CCT-ANK-11
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The project is terminated
Sponsor: Beijing Kejing Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCT-ANK-11
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumors (Pancreatic Cancer, Esophageal Cancer, Gastric Cancer, Cholangiocarcinoma, Lung Cancer and Ovarian Cancer)
MeSH Terms: conditions — Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Cholangiocarcinoma; Lung Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A group (Experimental)
  Interventions: Drug: Allogeneic NK（CCT-ANK-11)

INTERVENTIONS:
Drug: Allogeneic NK（CCT-ANK-11) — allogeneic natural killer cells

SUMMARY:
An exploratory clinical study to evaluate the safety and efficacy of NK cells (combined with standard therapy) in the treatment of solid tumor patients

ELIGIBILITY:
Inclusion Criteria:

1. The patient agrees to complete the entire treatment plan and sign the informed consent form.
2. Age 18 to 65, male or female.
3. Malignancy confirmed by histology or imaging diagnosis (computer tomography (CT), magnetic resonance imaging (MRI), contrast-enhanced ultrasound, EOB-MRI), the malignant solid tumor was completely resected (R0).
4. Patients who have received surgical treatment 4-8 weeks before the screening period.
5. Quality of life assessment form (ECOG) score 0,2.
6. Child-Pugh score of liver function ≤ 7.
7. The life expectancey is more than 6 months.
8. Patients with appropriate hematological functions:

（1）White blood cell (WBC) ≥ 3000 cells / mm3. （2）Absolute neutrophil count (ANC) ≥ 1500 cells.

（3）Platelet count (Platelets) ≥ 80000/mm3. （4）Hemoglobin (Hb) ≥ 9g/dl. 9. Patients with appropriate liver and kidney functions:

（1）Urea nitrogen (BUN) ≤ 1.5 times of the upper limit of normal value (ULN).（2）Serum creatinine (serumcreatinine) ≤ 1.5 times of the upper limit of normal value (ULN).（3）Total bilirubin (TB) ≤ 1.5 times of the upper limit of normal value (ULN).（4）Glutamic pyruvic transaminase (ALT or GPT) and glutamic oxaloacetic transaminase (AST or GOT) ≤ 2.5 times the upper limit of normal value (ULN).

10. Patients who have tested negative for syphilis and AIDS. 11.Patient with active hepatitis B, can take antiviral drugs during the trial period.

twelve。 Fertile men and women must use effective contraception within 14 days after signing the informed consent form and within 14 days after the last dose of natural killer cells are infused.

13. At least two forms of birth control must be used, one of which must be a barrier method. Acceptable contraceptive measures include:

（1）Establish oral, injection or implanted hormone contraceptive methods.（2）Placement of intrauterine device (IUD) or intrauterine system (IUS).（4）Barrier method: condom or occlusive cap (contraceptive diaphragm or cervical / uterine cap).

14. The patient agrees to comply to the trial rpotocols.

Exclusion Criteria:

1. Patients received drugs or other cellular immunotherapy in other clinical trials within 28 days before the screening period.
2. Patients are receiving immunosuppressive therapy for previous or recurrent autoimmune diseases within 14 days before allogeneic natural killer cell infusion.
3. The patient suffered from other malignant tumors in the past 5 years (except basal cell carcinoma or squamous cell carcinoma of the skin and carcinoma in situ of the cervix).
4. Acute illness in progress, or has been accompanied by serious diseases in the past 2 years, such as cardiovascular disease (such as New York Heart Association (NYHA) III or IV), mental health problems (e.g. alcohol, drug abuse). Or the program moderator judges patients who are not suitable to participate in clinical trials on the basis of medical history, physical examination results or test abnormalities that may interfere with the test results or adversely affect the safety of the subjects.
5. Allergic to aminoglycosides (Aminoglycoside) or subtilisin (Bacitracin), such as streptomycin (Streptomycin) and gentamicin (Gentamicin).
6. Patient is known to be allergic to any ingredient in the end product of NK preparation, including human serum albumin.
7. Female subjects who are breast-feeding or positive for serum or urine pregnancy tests during the screening period.
8. Pretreatment with steroids or antihistamines cannot be controlled for radiographic contrast agents (iodinated or non-iodinated) who have a history of allergy or allergic reactions or other clinically significant adverse reactions, and the researchers believe that it is not suitable for subjects who undergo conventional computerized tomography (CT) or magnetic resonance imaging (MRI). And subjects with contraindications for CT scanning for other reasons (such as strong magnetic implants, severe claustrophobia) should not be included in the group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and the efficacy | 12 months
  To evaluate the safety and objective remission rate of multiple injections of allogeneic natural killer cells (complete remission [CR] + partial remission [PR])

IPD SHARING:
Plan to Share IPD: No